CLINICAL TRIAL: NCT05984186
Title: Wingate-type Exercise Test to Evaluate the Effect of High Velocity Therapy on Recovery Sensation and Blood Lactate Decline
Brief Title: Effect of High Velocity/Hyperoxic Breathing Therapy on Blood Lactate Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: Auburn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RP-VTPF2022001Sci
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Dyspnea; Lactic Acidosis; Muscle; Breathlessness; Exercise; Recovery
MeSH Terms: conditions — Dyspnea; Acidosis, Lactic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- FiO2=100% with Flow=5LPM (Experimental): The study is a repeated measures model that will collect data on the participants with the designated HVT at four specified settings (Flow/FiO2) during the Wingate exercise test and during the recovery interval. The Wingate exercise test configuration, equipment and procedures will be repeated for each HVT setting for a matched dataset.
  The study will include four study arms, corresponding to four therapy settings being tested: (1) FiO2=100% with Flow=5LPM, (2) FiO2=21% with Flow=25-35LPM, (3) FiO2=100% with Flow=25-35LPM, (4) FiO2=21% with Flow=5LPM. The participants will wear the appropriately sized nasal cannula interface during the exercise and recovery.
  Interventions: Device: High Velocity Therapy
- FiO2=21% with Flow=25-35LPM (Experimental): The study is a repeated measures model that will collect data on the participants with the designated HVT at four specified settings (Flow/FiO2) during the Wingate exercise test and during the recovery interval. The Wingate exercise test configuration, equipment and procedures will be repeated for each HVT setting for a matched dataset.
  The study will include four study arms, corresponding to four therapy settings being tested: (1) FiO2=100% with Flow=5LPM, (2) FiO2=21% with Flow=25-35LPM, (3) FiO2=100% with Flow=25-35LPM, (4) FiO2=21% with Flow=5LPM. The participants will wear the appropriately sized nasal cannula interface during the exercise and recovery.
  Interventions: Device: High Velocity Therapy
- FiO2=100% with Flow=25-35LPM (Experimental): The study is a repeated measures model that will collect data on the participants with the designated HVT at four specified settings (Flow/FiO2) during the Wingate exercise test and during the recovery interval. The Wingate exercise test configuration, equipment and procedures will be repeated for each HVT setting for a matched dataset.
  The study will include four study arms, corresponding to four therapy settings being tested: (1) FiO2=100% with Flow=5LPM, (2) FiO2=21% with Flow=25-35LPM, (3) FiO2=100% with Flow=25-35LPM, (4) FiO2=21% with Flow=5LPM. The participants will wear the appropriately sized nasal cannula interface during the exercise and recovery.
  Interventions: Device: High Velocity Therapy
- FiO2=21% with Flow=5LPM (Experimental): The study is a repeated measures model that will collect data on the participants with the designated HVT at four specified settings (Flow/FiO2) during the Wingate exercise test and during the recovery interval. The Wingate exercise test configuration, equipment and procedures will be repeated for each HVT setting for a matched dataset.
  The study will include four study arms, corresponding to four therapy settings being tested: (1) FiO2=100% with Flow=5LPM, (2) FiO2=21% with Flow=25-35LPM, (3) FiO2=100% with Flow=25-35LPM, (4) FiO2=21% with Flow=5LPM. The participants will wear the appropriately sized nasal cannula interface during the exercise and recovery.
  Interventions: Device: High Velocity Therapy

INTERVENTIONS:
Device: High Velocity Therapy — FiO2=100% with Flow=5LPM FiO2=21% with Flow=25-35LPM FiO2=100% with Flow=25-35LPM FiO2=21% with Flow=5LPM

SUMMARY:
The study will evaluate the impact of high velocity therapy (HVT) on reduction of work of breathing (as implied by breath frequency) and enhanced blood lactate decline during recovery from a Wingate-type Exercise test. The study will include four study segments, corresponding to four different therapy settings.

DETAILED DESCRIPTION:
HVT has been found to be a useful clinical tool for treatment of Type 1 and Type 2 respiratory failure (including hypercapnic respiratory failure), acute decompensated heart failure, and COVID respiratory complications. The overall objective of this prospective, pilot study is to evaluate whether HVT might enhance the decline of blood lactate concentrations following a high intensity exercise bout, in healthy volunteers. The hypothesis is that HVT, regardless of the oxygen concentration (i.e., FiO2), will reduce the work of breathing and increase the lactate clearance rate during exercise and recovery intervals. This pilot study could ignite further research providing HVT applications to high performing athletics and patients in an acute care setting requiring physical rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults18-30 years old, in a general state of good health, of either sex
* No known contraindication to performing a maximal exercise test, i.e., Wingate-type Anaerobic exercise test
* Participants must consider themselves able to perform "regular moderate" or "regular strenuous" exercise.
* ° "Regular moderate" exercise includes less than 30 minutes every day or 30 minutes every other day, of some form of deliberate exercise, that does not include walking.
* ° "Regular strenuous" exercise is 30+ minutes per day, of some form of deliberate exercise, that does not include walking.

Exclusion Criteria:

* Not considered a 'high-performance athlete'
* Known active cardiovascular, metabolic, liver, or renal disease
* Orthopedic limitations to exercise
* Pregnancy
* Use of beta-blockers or beta-agonist asthma medications
* Exercise induced asthma
* Any other health-related issue that would involve the participant's fitness capability
* Inability to complete all of the study procedures

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Gladden, Principal Investigator — Auburn University; Michael Roberts, Principal Investigator — Auburn University; Max Michael, Principal Investigator — Auburn University; Nina Stute, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Subjects will receive High Velocity Therapy. There will be four different flow settings and FIO2 for a total of four groups. Each participants will complete all four arms in randomized order.
  All 15 patients completed all 4 arms.
  FiO2=100% with Flow=5LPM FiO2=21% with Flow=25-35LPM FiO2=100% with Flow=25-35LPM FiO2=21% with Flow=5LPM
Period: FiO2=100% With Flow=5LPM
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: FiO2=21% With Flow=25-35LPM
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: FiO2=100% With Flow=25-35LPM
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: FiO2=21% With Flow=5LPM
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subject will receive High Velocity Therapy; four different flow settings and FIO2 for a total of four groups.
  FiO2=100% with Flow=5LPM FiO2=21% with Flow=25-30LPM FiO2=100% with Flow=25-30LPM FiO2=21% with Flow=5LPM
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Blood Lactate Change
Description: The change in blood lactate starting from the exercise test throughout the recovery period
Time Frame: At rest (TR) and during recovery from the Wingate test at minute 2 (T2) minute 4 (T4), minute 6 (T6), minute 8 (T8), minute 10 (T10) minute 15 (T15), minute 20 (T20), minute 25 (T25), minute 30 (T30) minute 40 (T40), minute 50 (T50) minute 60 (T60).
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- FiO2=21% With Flow=5LPM; FiO2=21% With Flow=25-35LPM; FiO2=100% With Flow=5LPM; FiO2=100% With Flow=25-35LPM: High Velocity Therapy: Four different flow settings and FiO2
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
mmol/L
  TR | 1.19 (.49) | 1.22 (.98) | 1.11 (.36) | 1.05 (.42)
  T2 | 9.85 (2.24) | 9.63 (2.32) | 9.55 (1.48) | 9.56 (2.19)
  T4 | 11.05 (2.16) | 10.75 (2.24) | 10.86 (1.90) | 10.61 (2.19)
  T6 | 11.60 (1.96) | 11.33 (2.03) | 10.83 (1.81) | 10.89 (2.05)
  T8 | 11.30 (2.22) | 11.29 (2.49) | 11.14 (1.96) | 10.26 (1.91)
  T10 | 11.30 (2.33) | 11.13 (2.41) | 10.63 (2.03) | 10.22 (1.92)
  T15 | 10.07 (2.36) | 9.59 (2.42) | 9.43 (2.01) | 9.16 (2.37)
  T20 | 8.73 (2.24) | 8.20 (2.26) | 8.04 (2.06) | 7.73 (2.02)
  T25 | 7.39 (2.14) | 6.90 (2.03) | 6.72 (1.99) | 6.53 (1.91)
  T30 | 6.22 (1.66) | 5.84 (1.91) | 5.49 (1.52) | 5.47 (1.63)
  T40 | 4.49 (1.29) | 4.31 (1.59) | 4.07 (1.23) | 3.99 (1.21)
  T50 | 3.39 (.95) | 3.27 (1.10) | 2.95 (.91) | 2.96 (.94)
  T60 | 2.26 (.73) | 2.61 (.90) | 2.37 (.72) | 2.41 (.73)

2. Secondary Outcome: Respiratory Rate Change
Description: The change in respiratory rate starting from the exercise test throughout the recovery period
Time Frame: Prior to the Wingate test (TR) and after at 1min (T1), 2min (T2), 4min (T4), 6min (T6), 8min (T8), 10min (T10), 15min (T15), 20min (T20), 25min (T25), 30min (T30), 40min (T40), 50 min (T50), and 60min (T60) into recovery.
Population: Subjects that had the data collected for the specified time point.
Measure: Mean (Standard Deviation); unit: Breaths per min
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
Breaths per min
  TR: number analyzed (Participants) | 15 | 14 | 15 | 15
  TR | 14.04 (4.71) | 14.35 (3.91) | 15.24 (5.93) | 13.59 (3.79)
  T1: number analyzed (Participants) | 14 | 13 | 15 | 15
  T1 | 29.01 (5.19) | 25.05 (7.34) | 25.41 (8.02) | 27.3 (5.53)
  T2 | 25.63 (6.81) | 25.97 (5.45) | 25.59 (6.02) | 22.73 (6.52)
  T4 | 25.53 (5.95) | 22.47 (6.85) | 22.63 (6.67) | 21.39 (6.29)
  T6 | 22.98 (5.81) | 20.18 (5.97) | 20.04 (7.25) | 19.09 (5.83)
  T8 | 20.33 (6.84) | 18.04 (4.78) | 19.02 (8.39) | 17.84 (6.80)
  T10 | 21.20 (4.19) | 18.91 (4.20) | 18.35 (6.45) | 17.51 (5.72)
  T15 | 19.12 (5.17) | 16.19 (3.91) | 17.91 (5.31) | 15.17 (7.04)
  T20 | 17.89 (5.56) | 14.05 (3.61) | 16.51 (6.58) | 14.32 (5.54)
  T25 | 16.20 (5.90) | 12.64 (4.40) | 16.61 (5.07) | 13.07 (4.90)
  T30 | 16.01 (4.66) | 12.00 (5.05) | 12.91 (4.45) | 12.68 (4.56)
  T40 | 15.09 (4.82) | 11.59 (3.01) | 12.92 (4.31) | 12.46 (4.68)
  T50 | 14.03 (4.19) | 11.43 (3.83) | 13.14 (6.73) | 10.81 (3.94)
  T60 | 14.03 (3.24) | 10.77 (3.64) | 12.99 (4.85) | 10.83 (2.86)

3. Secondary Outcome: Heart Rate Change
Description: The change in heart rate starting from the exercise test throughout the recovery period
Time Frame: Prior to the Wingate test (TR) and after 2min (T2), 4min (T4), 6min (T6), 8min (T8), 10min (T10), 15min (T15), 20min (T20), 25min (T25), 30min (T30), 40min (T40), 50 min (T50), and 60min (T60) into recovery.
Population: Subjects that had this data collected for the specified time point.
Measure: Mean (Standard Deviation); unit: Beats per min
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
Beats per min
  TR: number analyzed (Participants) | 15 | 14 | 15 | 15
  TR | 78.7 (11.87) | 77.43 (10.93) | 77.33 (11.08) | 81.13 (14.94)
  T2 | 121.60 (10.03) | 120.53 (17.22) | 117.13 (7.64) | 116.93 (12.14)
  T4 | 107.27 (10.98) | 107.93 (11.97) | 103.27 (10.40) | 105.00 (10.45)
  T6 | 103.33 (8.59) | 106.27 (11.65) | 100.80 (10.36) | 101.20 (9.95)
  T8 | 102.93 (8.53) | 104.67 (10.76) | 101.73 (8.55) | 101.20 (9.12)
  T10 | 100.73 (8.83) | 102.73 (10.50) | 101.80 (10.18) | 99.87 (8.36)
  T15 | 98.73 (8.96) | 101.00 (7.65) | 97.86 (7.85) | 97.20 (10.48)
  T20 | 97.13 (9.49) | 98.47 (8.40) | 95.80 (9.37) | 95.13 (10.23)
  T25 | 96.87 (11.11) | 96.27 (10.93) | 93.20 (9.26) | 93.33 (10.44)
  T30 | 93.40 (10.18) | 95.93 (9.91) | 94.80 (9.21) | 94.07 (9.48)
  T40 | 93.87 (11.18) | 90.53 (8.72) | 92.47 (8.43) | 89.47 (9.58)
  T50 | 90.73 (8.25) | 90.53 (9.35) | 89.00 (9.89) | 90.00 (12.26)
  T60 | 89.47 (8.90) | 89.87 (10.79) | 85.57 (9.00) | 86.13 (9.31)

4. Secondary Outcome: SpO2 Change
Description: The change in SpO2 starting from the exercise test throughout the recovery period.
Time Frame: Prior to the Wingate test (TR) and after at, 2min (T2), 4min (T4), 6min (T6), 8min (T8), 10min (T10), 15min (T15), 20min (T20), 25min (T25), 30min (T30), 40min (T40), 50 min (T50), and 60min (T60) into recovery.
Population: Subjects that had the data collected at that specified time point.
Measure: Mean (Standard Deviation); unit: Percent oxygen
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
Percent oxygen
  TR: number analyzed (Participants) | 15 | 14 | 15 | 15
  TR | 99.07 (.80) | 98.71 (1.14) | 98.13 (1.60) | 98.49 (.99)
  T2 | 98.20 (.94) | 98.13 (1.13) | 98.47 (1.46) | 99.33 (.72)
  T4 | 97.73 (1.10) | 97.53 (1.13) | 98.53 (.83) | 99.00 (.85)
  T6 | 97.73 (.96) | 96.80 (1.52) | 98.27 (1.10) | 99.00 (.85)
  T8 | 97.00 (1.31) | 96.87 (.99) | 98.33 (.90) | 98.87 (.64)
  T10 | 97.20 (1.08) | 96.60 (.83) | 98.27 (.88) | 98.47 (1.46)
  T15 | 96.87 (.99) | 96.33 (.90) | 98.13 (.74) | 98.27 (1.33)
  T20: number analyzed (Participants) | 15 | 14 | 15 | 15
  T20 | 96.53 (1.06) | 96.43 (.94) | 98.13 (.74) | 98.47 (.74)
  T25 | 96.47 (1.19) | 95.87 (1.55) | 98.00 (.76) | 98.00 (1.41)
  T30 | 95.80 (1.15) | 96.00 (1.20) | 97.73 (.96) | 98.27 (.96)
  T40 | 96.00 (1.89) | 95.73 (1.22) | 98.87 (.64) | 97.60 (2.38)
  T50 | 96.00 (1.20) | 96.27 (1.33) | 98.13 (.64) | 98.00 (1.89)
  T60 | 96.00 (1.41) | 95.87 (1.41) | 97.71 (.73) | 98.07 (2.37)

5. Secondary Outcome: Systolic Blood Pressure Change
Description: The change in systolic blood pressure starting from the exercise test throughout the recovery period.
Time Frame: Prior to the Wingate test (TR) and after at, 5min (T5) 10min (T10), 15min (T15), 20min (T20), 25min (T25), 30min (T30), 40min (T40), 50 min (T50), and 60min (T60) into recovery.
Population: Subjects that had this data collected for the specified time point.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
mmHG
  TR | 125.73 (16.88) | 126.27 (8.49) | 125.20 (12.40) | 121.33 (10.47)
  T5: number analyzed (Participants) | 15 | 14 | 15 | 15
  T5 | 132.87 (17.11) | 138.57 (20.49) | 136.53 (16.25) | 133.93 (13.60)
  T10: number analyzed (Participants) | 14 | 15 | 15 | 15
  T10 | 124.14 (15.03) | 123.47 (13.94) | 126.47 (12.72) | 125.20 (15.84)
  T15: number analyzed (Participants) | 13 | 14 | 14 | 15
  T15 | 124.31 (15.48) | 120.93 (13.79) | 124.86 (13.20) | 124.46 (12.76)
  T20: number analyzed (Participants) | 15 | 14 | 15 | 15
  T20 | 117.93 (17.26) | 118.93 (13.65) | 120.80 (15.79) | 120.79 (15.49)
  T25: number analyzed (Participants) | 15 | 14 | 15 | 15
  T25 | 116.60 (14.27) | 117.86 (10.74) | 114.20 (10.69) | 115.07 (13.37)
  T30 | 115.40 (12.07) | 116.67 (10.19) | 116.87 (13.33) | 114.07 (14.03)
  T40 | 114.33 (14.94) | 114.93 (11.16) | 116.60 (12.89) | 113.93 (8.34)
  T50 | 117.47 (21.23) | 114.47 (9.77) | 115.87 (10.49) | 1113.93 (11.32)
  T60: number analyzed (Participants) | 14 | 15 | 15 | 15
  T60 | 114.07 (12.46) | 114.47 (11.12) | 114.86 (9.43) | 113.67 (11.31)

6. Secondary Outcome: Diastolic Blood Pressure Change
Description: The change in diastolic blood pressure change starting from the exercise test throughout the recovery period.
Time Frame: as for outcome 5
Population: Subjects that had this data collected for the specified time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
mmHg
  TR | 75.73 (8.50) | 76.73 (7.86) | 75.53 (8.56) | 75.00 (9.46)
  T5: number analyzed (Participants) | 15 | 14 | 15 | 15
  T5 | 67.20 (8.60) | 69.14 (8.96) | 68.93 (5.64) | 68.53 (6.72)
  T10: number analyzed (Participants) | 14 | 15 | 15 | 15
  T10 | 70.00 (10.99) | 70.20 (6.67) | 69.40 (4.55) | 72.20 (16.40)
  T15: number analyzed (Participants) | 13 | 15 | 14 | 15
  T15 | 71.31 (14.33) | 70.80 (12.19) | 74.29 (5.46) | 69.92 (6.63)
  T20: number analyzed (Participants) | 15 | 14 | 15 | 15
  T20 | 70.47 (6.06) | 72.57 (7.24) | 77.67 (20.70) | 77.07 (18.85)
  T25: number analyzed (Participants) | 15 | 14 | 15 | 15
  T25 | 70.27 (6.60) | 74.86 (9.45) | 70.53 (6.14) | 74.07 (11.15)
  T30 | 70.13 (7.18) | 72.07 (7.08) | 69.93 (4.68) | 70.87 (8.84)
  T40 | 69.27 (9.09) | 76.60 (12.48) | 72.80 (11.45) | 76.13 (12.86)
  T50 | 72.27 (20.09) | 71.27 (7.64) | 71.07 (6.61) | 71.73 (7.27)
  T60: number analyzed (Participants) | 14 | 15 | 15 | 15
  T60 | 69.71 (7.72) | 71.40 (9.16) | 71.50 (5.23) | 71.33 (5.75)

7. Secondary Outcome: Perceived Level of Exertion Change
Description: The change in the subjects perceived level of exertion starting from after the exercise test throughout the recovery period. The scale will be 0-10; a lower score is a lower level of exhaustion, a higher score is a higher level of exhaustion.
Time Frame: Immediately after the Wingate test (T0) and after at, 2min (T2), 4min (T4), 6min (T6), 8min (T8), 10min (T10), 15min (T15), 20min (T20), 25min (T25), 30min (T30), 40min (T40), 50 min (T50), and 60min (T60) into recovery.
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | FiO2=21% With Flow=5LPM | FiO2=21% With Flow=25-35LPM | FiO2=100% With Flow=5LPM | FiO2=100% With Flow=25-35LPM
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale (0-10)
  T0 | 8.40 (2.10) | 7.86 (2.80) | 8.54 (1.98) | 8.93 (1.33)
  T2 | 7.07 (1.87) | 6.87 (2.47) | 6.93 (2.02) | 6.93 (1.75)
  T4 | 5.73 (2.25) | 5.87 (2.50) | 5.67 (2.13) | 5.80 (1.47)
  T6 | 4.80 (2.34) | 4.93 (2.71) | 5.00 (2.20) | 4.60 (1.68)
  T8 | 4.13 (2.07) | 4.13 (2.75) | 3.87 (2.45) | 3.67 (2.29)
  T10 | 3.67 (2.32) | 3.67 (2.53) | 3.47 (2.61) | 3.07 (2.19)
  T15 | 2.80 (2.18) | 2.67 (2.19) | 2.60 (2.13) | 2.47 (2.07)
  T20 | 2.33 (2.06) | 2.27 (2.12) | 2.20 (1.90) | 2.07 (1.79)
  T25 | 2.07 (1.94) | 1.93 (1.87) | 1.80 (1.78) | 1.67 (1.54)
  T30 | 1.73 (1.62) | 1.47 (1.64) | 1.67 (1.68) | 1.43 (1.55)
  T40 | 1.40 (1.35) | 1.27 (1.49) | 1.13 (1.36) | 1.13 (1.19)
  T50 | .93 (.96) | .93 (1.03) | .93 (1.03) | 1.07 (1.22)
  T60 | .73 (.80) | .60 (.74) | .71 (.73) | .93 (.96)

ADVERSE EVENTS:
Time Frame: The starting point was the exercise test, and AE data was collected throughout the recovery period for a total of 60 min. This was repeated for each arm, on different days.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- All Participants: Subject will receive High Velocity Therapy; four different flow settings and FIO2 for a total of four groups.
  FiO2=100% with Flow=5LPM FiO2=21% with Flow=25-35LPM FiO2=100% with Flow=25-35LPM FiO2=21% with Flow=5LPM
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT05984186/Prot_SAP_000.pdf